CLINICAL TRIAL: NCT01327170
Title: Micropulse Diode Laser Treatment for Chronic Central Serous Chorioretinopathy: Evaluation by Fundus Autofluorescence and Spectral Domain Optical Coherence Tomography
Brief Title: Micropulse Diode Laser Treatment for Chronic Central Serous Chorioretinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Fernanda Pedreira Magalhães, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDMCCSC-FM
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Central Serous Chorioretinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subthreshold diode micropulse laser (Active Comparator): Subthreshold diode micropulse laser in patients with chronic central serous chorioretinopathy
  Interventions: Procedure: Subthreshold diode micropulse laser
- Sham (Sham Comparator): Sham group simulating the laser treatment
  Interventions: Procedure: Subthreshold diode micropulse laser

INTERVENTIONS:
Procedure: Subthreshold diode micropulse laser

SUMMARY:
The aim of this study was to evaluate safety and therapeutic response to micropulse diode 810nm laser treatment in patients with chronic central serous chorioretinopathy.

DETAILED DESCRIPTION:
Most of the cases of central serous chorioretinopathy (CSC) recur spontaneously within three months of disease. After 3 months without resolution of acute CSC or in chronic CSC, continuous wave laser photocoagulation or photodynamic therapy should be considered. Direct threshold continuous photocoagulation treatment can shorten the duration of the serous detachment, but it is not appropriate for juxtafoveal or subfoveal leakage point.Subvisible photocoagulation potentially localizes and decreases chorioretinal thermic burn. Subthreshold diode micropulse (SDM) laser using a 810nm diode laser may spare the damage to the neural retina by raising the temperature of the RPE to just below the protein-denaturation threshold so that the thermal wave that reaches the neural retina is insufficient to cause neither damage nor clinically visible end-point. This therapeutic laser modality offers the possibility to minimize the iatrogenic retinal lesion.

ELIGIBILITY:
Inclusion Criteria:

* Chronic active central serous chorioretinopathy lasting more than 6 months
* Leakage at fluorescein angiogram

Exclusion Criteria:

* Opacities of the clear refractive media of the eye
* Any intraocular surgery within the 6 months prior to study entry
* Prior vitrectomy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 6 months
  Best corrected visual acuity measured by ETDRS chart at baseline, 1, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Macular subretinal fluid | 6 months
  Central macular thickness measured by spectral-domain optical coherence tomography at baseline, 1, 3, 6, 9 and 12 months
Leakage at fluorescein angiogram | 6 months
  Leakage at fluorescein angiogram evaluated at baseline, 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda P Magalhaes, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203